CLINICAL TRIAL: NCT00306839
Title: Prospective, Controlled, Randomized Study to Evaluate Pain and Further Disabling Complications in Patients Undergoing Lichtenstein Technique for Primary Inguinal Hernia Repair by Fixing the Mesh With Fibrin Sealant Versus Sutures
Brief Title: Efficacy Study of Tissucol/Tisseel Fibrin Sealant to Treat Inguinal Hernia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Milan (Other)
Collaborators: Baxter Healthcare Corporation (Industry); Pr Giampiero CAMPANELLI (Unknown)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TIMELI 001
Record Dates: First submitted 2006-03-22; First posted 2006-03-24 (Estimated); Last update posted 2009-02-13 (Estimated); Status verified 2009-02

CONDITIONS: Inguinal Hernia
Keywords: Tissucol; Tisseel; Lichtenstein; hernia; inguinal
MeSH Terms: conditions — Hernia, Inguinal; Hernia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Other): Tissel group
  Interventions: Procedure: standardized Lichtenstein technique
- 2 (Other): Suture group
  Interventions: Procedure: standardized Lichtenstein technique

INTERVENTIONS:
Procedure: standardized Lichtenstein technique

SUMMARY:
The purpose of the study is to evaluate mid and long term postoperative pain and further disabling complications in open inguinal hernia repair by Lichtenstein technique after mesh fixation with fibrin sealant (FS), compared to mesh fixation with sutures.

DETAILED DESCRIPTION:
Subjects in the FS group will be operated by Lichtenstein technique, with mesh fixation by fibrin sealant. Subjects in control group will be operated with conventional Lichtenstein technique (mesh fixation by sutures).

Hernia repair will be performed according to standardized Lichtenstein technique, a technique for tension free hernioplasty. A Polypropylene, heavyweight, macroporous mesh will be used (8x15 cm) tailored to individual patients requirement. The different ways of mesh fixation will be randomly assigned within 24 hours before the operation. In the FS group, the two tails of the mesh will be fixed together in overlapping their edges and by surrounding the cord. The edges will be joined up to by 1 suture. No other sutures will be used. First the mesh will be put correctly in place. A small spot (0.5ml) of FS will be applied on the pubis under the mesh without spray then the remaining part (3,5ml) over the mesh on the entire surface in a thin uniform layer by spray. 2 ml Tissucol-Tisseel (4 ml of fibrin sealant) will be used per mesh. In the control group, the mesh will be fixed in a conventional manner. Nerve resection (if occurred) will be recorded; it should be avoided.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent obtained from the subject prior to participation in the study
* Active males over the age of 18 years and below 80 years
* Experiencing an uncomplicated unilateral primary inguinal hernia or experiencing an uncomplicated bilateral hernia provided that only one hernia is operated during the 12 months of study follow-up
* Subjects eligible for elective inguinal hernia repair using Lichtenstein technique.

Exclusion Criteria:

* Recurrent, scrotal, incarcerated or femoral hernias
* Hernia types L3 and M3 according the EHS classification
* BMI equal or more than 35
* Concomitant abdominal surgery
* Ongoing long term analgesic or steroid treatment
* Patients under Clopidogrel or Warfarin (can be switched to LMW sub-cutaneous heparin)
* Known abuse of alcohol or drugs
* Liver cirrhosis (Child C)
* Previous treatment or Hypersensitivity to bovine aprotinin
* Known immunodeficiency
* Severely compromised physical or psychological health, that in the investigator's opinion will affect patient compliance
* Concurrently participating in another clinical trial and having received another investigational drug or device within the last 30 days

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 325 (Actual)
Dates: Start 2006-02; Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Combined endpoint evaluating incidence of disabling complications:chronic pain and/or numbness and/or groin discomfort assessed 1 year after surgery.

SECONDARY OUTCOMES:
Recurrence
Overall wound-healing complication rate (bleeding complications, bruising, seroma, wound infection, mesh infection)
Early postoperative pain at W1 and M1
Mid-term postoperative pain at M6
Incidence of patients without pain at M1, M6 and M12
Use of analgesic drugs
Patient's satisfaction
Safety (incidence of adverse events)
Quality of Life assessed by SF12 pre-operatively or at D-1, M1, M6 and M12
Hospital stay (hour or Days) and time to return to normal activities
A subgroup analysis will be done for patients receiving pre-operatively aspirin or LMW sub-cutaneous heparin.
The study will be blinded for the patient and for the physician evaluating the pain.

CONTACTS AND LOCATIONS:
Overall Officials: CAMPANELLI Giampiero, Professor, Study Chair
Locations (6):
- Gasthuisberg University Hospitals KUL, Leuven, Belgium
- Copenhagen university hospital, Gentofte, Hellerup, Denmark
- Hôpital Jean Verdier, Bondy, France
- St. Hildegardis-Krankenhaus, Mainz, Germany
- Clinica Nuestra Senora del Rosario, Madrid, Spain
- Derriford Hospital, Plymouth, United Kingdom

REFERENCES:
- [Derived] Campanelli G, Pascual MH, Hoeferlin A, Rosenberg J, Champault G, Kingsnorth A, Miserez M. Randomized, controlled, blinded trial of Tisseel/Tissucol for mesh fixation in patients undergoing Lichtenstein technique for primary inguinal hernia repair: results of the TIMELI trial. Ann Surg. 2012 Apr;255(4):650-7. doi: 10.1097/SLA.0b013e31824b32bf. PMID 22395092